CLINICAL TRIAL: NCT06621563
Title: Safety, Tolerability, Efficacy, Pharmacokinetics Profile and Immunogenicity of HS-20117 in Combination With Other Drugs in Advanced Solid Tumors, a Phase Ib Clinical Trial
Brief Title: Phase Ib Trial of HS-20117 in Combination With Other Drugs in Advanced Solid Tumors
Acronym: HS-20117
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Hansoh BioMedical R&D Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: HS-20117-102
Record Dates: First submitted 2024-09-29; First posted 2024-10-01 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Solid Tumors; Non-Small Cell Lung Cancer; Colorectal Cancer
Keywords: Solid tumor; EGFR/c-MET bispecific antibody; B7H3 ADC; chemotherapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Colorectal Neoplasms | interventions — Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (6):
- Cohort 1a (Experimental): NSCLC
  Interventions: Drug: HS-20117 combined Platinum-containing chemotherapy
- Cohort 2a (Experimental): NSCLC
  Interventions: Drug: HS-20117 combined HS-20093
- Cohort 3a (Experimental): CRC
  Interventions: Drug: HS-20117+CAPEOX
- Cohort 4a (Experimental): CRC
  Interventions: Drug: HS-20117+FOLFIRI
- Cohort 5a (Experimental): CRC
  Interventions: Drug: HS-20117+mFOLFOX6
- Cohort 6a (Experimental): CRC
  Interventions: Drug: HS-20117 combined HS-20093 and 5-FU

INTERVENTIONS:
Drug: HS-20117 combined HS-20093 — HS-20117 + HS-20093
  Arms: Cohort 2a
Drug: HS-20117 combined Platinum-containing chemotherapy — HS-20117 + cisplatin/carboplatin + pemetrexed
  Arms: Cohort 1a
Drug: HS-20117 combined HS-20093 and 5-FU — HS-20117 + HS-20093 + 5-FU
  Arms: Cohort 6a
Drug: HS-20117+CAPEOX — CAPOEX: Oxaliplatin+Capecitabine
  Arms: Cohort 3a
Drug: HS-20117+FOLFIRI — FOLFIRI=Irinotecan+Leucovorin Calcium+5-FU
  Arms: Cohort 4a
Drug: HS-20117+mFOLFOX6 — mFOLFOX6=Oxaliplatin+Leucovorin Calcium+5-FU
  Arms: Cohort 5a

SUMMARY:
HS-20117 is a fully-human EGFR-MET immunoglobulin G1(IgG1)-like bispecific antibody. The purpose of study is to evaluate the safety, tolerability, efficacy, PK profile and immunogenicity of HS-20117 in combination with other drugs in advanced solid tumors.

DETAILED DESCRIPTION:
This is a multicenter, open-label, Phase Ib clinical trial of HS-20117 combination therapies to evaluate the safety, tolerability, efficacy, PK profile and immunogenicity in participants with advanced solid tumors. The study includes a dose escalation part and a dose expansion part. The dose-escalation study will be performed to evaluate the safety, tolerability, PK profile, immunogenicity, and efficacy of HS-20117 combination therapies in participants with advanced solid tumor. The subsequent dose-expansion study will be performed to evaluate the efficacy of HS-20117 combination therapies in participants with locally advanced or metastatic NSCLC harboring EGFR exon 20 insertion mutations or EGFR classical mutations, and RAS/BRAF V600E wild type CRC.

ELIGIBILITY:
Inclusion Criteria:

* Males or females aged 18 - 75 years (inclusive).
* Histologically confirmed unresectable, recurrent or metastatic solid tumors.
* At least one target lesion per the RECIST v1.1.
* ECOG performance status of 0-1.
* Minimum life expectancy > 12 weeks.
* Males or Females should be using adequate contraceptive measures throughout the study.
* Females must not be pregnant at screening or have evidence of non-childbearing potential.
* Signed Informed Consent Form.

Exclusion Criteria:

* Received or are receiving the following treatments:

  1. Any anticancer therapy targeting MET, including TKIs, antibodies or antibody-drug conjugates.
  2. Monoclonalor bispecific antibodies targeting EGFR.
  3. Systemic anti-cancer treatment (Cytotoxicities and anti-cancer Traditional Chinese medicine or TKIs) within 2 weeks prior to the first dose of HS-20117.
  4. Investigational anti-cancer drugs or antibodies or ADCs within 4 weeks prior to the first dose of HS-20117.
  5. Local radiotherapy within 2 weeks prior to the first dose of HS-20117, more than 30% of bone marrow irradiation or large-area radiotherapy within 4 weeks before the first dose of HS-20117.
  6. Presence of pleural effusion/ascites requiring clinical intervention; presence of pericardial effusion.
  7. Major surgery within 4 weeks prior to the first dose of HS-20117.
* Presence of Grade ≥ 2 toxicities due to prior anti-tumor therapy.
* Presence of uncured secondary primary malignancies.
* Untreated, or active central nervous system metastases.
* Severe, uncontrolled or active cardiovascular disorders.
* Serious infection within 4 weeks prior to the first dose of HS-20117.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 780 (Estimated)
Dates: Start 2024-12-14 (Actual); Primary Completion 2026-03-30 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of treatment-emergent adverse events | rom the date of first dose to 90 days after the final dose.
  Adverse event (assessed according to NCI CTCAE v5.0) is defined as any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship.
Tolerability of HS-20117 combination therapy: incidence of DLT events, maximum tolerated dose (MTD) or maximum applicable dose (MAD) of HS-20117 in combination therapies. | From the date of first dose to day 21.
  MTD is defined as the previous dose level at which 2 or more out of 2-6 subjects experienced a DLT. MAD is defined as follows: a) based on PK data, it is anticipated that at this dose level, the dose-exposure plateau has been reached, b) based on existing safety data, it is judged that dose escalation following this dose level will have a large safety risk or subject intolerance, or c) based on the PK-PD model, it suggested that the optimal target concentration of safety and efficacy has been explored.

SECONDARY OUTCOMES:
Efficacy of HS-20117: Objective response rate (ORR) | From the date of first dose to the date of disease progression or withdrawal from study, approximately 2 years
  ORR is defined as the percentage of participants with BOR of confirmed CR or confirmed PR per RECIST v1.1
Efficacy of HS-20117: disease control rate (DCR) | From the date of first dose to the date of disease progression or withdrawal from study, approximately 2 years
  DCR is deﬁned as the percentage of patients who have a best overall response (confirmed CR, PR, or stable disease for at least 6 weeks) per RECIST v1.1.
Efficacy of HS-20117: duration of response (DoR) | From the date of first dose to the date of disease progression or withdrawal from study, approximately 2 years
  DoR only applies to participants whose best overall response is CR or PR based on assessment per RECIST v1.1. The start date is the date of first documented response of CR or PR (i.e. the start date of observed response, not the date when response was confirmed), and the end date is defined as the date of the first documented progression or death due to underlying disease.
Efficacy of HS-20117: progression free survival (PFS) | From the date of first dose to the date of disease progression or withdrawal from study, approximately 2 years
  PFS is defined as the time from the date of randomization or first dose (if randomization is not needed) to the date of the first documented progression or death due to any cause. PFS will be assessed per RECIST v1.1.
Efficacy of HS-20117: overall survival (OS) | From the date of first dose to the date of disease progression or withdrawal from study, approximately 2 years
  OS is defined as the time from the date of randomization or first dose (if randomization is not needed) to the date of death due to any cause. For each participant who is not known to have died as of the cutoff date for overall survival analysis, OS time was censored on the last date the participant is known to be alive.
PK parameters: Trough serum concentration (Ctrough) of HS-20117 and HS-20093 | From the date of first dose to 90 days after the final dose.
  Ctrough is the observed serum concentration immediately prior to the next administration.
PK parameters: Time to reach maximum observed serum concentration (Tmax) of HS-20117 | From the date of first dose to 90 days after the final dose.
  The Tmax is defined as time to reach maximum observed serum concentration of HS-20117.
PK parameters: Area under the curve from time Zero to end of dosing interval (AUCtau) of HS-20117 | From the date of first dose to 90 days after the final dose.
  The AUCtau is defined as the area under the serum concentration-time curve during a dose interval time period (tau).
PK parameters: Maximum serum concentration (Cmax) of HS-20117 and HS-20093. | From the date of first dose to 90 days after the final dose.
  The Cmax is the maximum observed serum concentration of HS-20117, HS-20093.
Immunogenicity of HS-20117 | From the date of first dose to 90 days after the final dose.
  Immunogenicity will be measured by the number of participants that are ADA positive.

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Medical University Cancer Institute & Hospital, Tianjin, China

IPD SHARING:
Plan to Share IPD: No